CLINICAL TRIAL: NCT05702918
Title: Evaluation of the Course and Effectiveness of Conservative Therapy in Patients With Achilles Tendinopathy Using Ultrasonography
Brief Title: Evaluation of the Course and Effectiveness of Conservative Therapy in Patients With Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Stanislav Machač, Ph.D, Academic worker, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK-402 /22
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2023-12

CONDITIONS: Achilles Tendinopathy
Keywords: Achilles Tendinopathy; Extracorporeal Shockwave Therapy; Ultrasonography

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups. Group A will follow resistance training protocol and receive ESWT. Group B will follow resistance training only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - ESWT + exercise (Active Comparator): Participants in group A will complete a 12-week ankle dorsiflexion resistance training protocol according to Silbernagel. It is a series of heel rise exercises with a gradual progression of load according to defined criteria, which the patient practices every day.
  In addition, participants will receive a low-energy focused ESWT. In total, it will be applied 4 times with an interval of 7 days from the BTL-6000 FSWT device with piezoelectric generator. The energy will be set to 0.10-0.14 mJ/mm2, frequency 5 Hz, total number of shocks 2000. The application will be semi-static at the location of the largest USG finding. Shocks are applied from all three sides (medial, lateral, dorsal). The set values will not change throughout the research. These parameters were selected in accordance to ISMST guidelines.
  Interventions: Device: BTL-6000 FSWT; Other: Achilles Tendon Loading Exercise Protocol According to Silbernagel
- Group B - exercise (Active Comparator): Participants in group B will complete a 12-week ankle dorsiflexion resistance training protocol according to Silbernagel. It is a series of heel rise exercises with a gradual progression of load according to defined criteria, which the patient practices every day.
  Interventions: Other: Achilles Tendon Loading Exercise Protocol According to Silbernagel

INTERVENTIONS:
Device: BTL-6000 FSWT — The energy will be set to 0.10-0.14 mJ/mm2, frequency 5 Hz, total number of shocks 2000. The application will be semi-static at the location of the largest USG finding. Shocks are applied from all three sides (medial, lateral, dorsal).
  Arms: Group A - ESWT + exercise
Other: Achilles Tendon Loading Exercise Protocol According to Silbernagel — It is a 12-week Silbernagel ankle dorsiflexion resistance training protocol. It is a series of exercises with a gradual progression of load according to defined criteria, which the patient practices every day.

SUMMARY:
This work is designed as a randomized clinical trial, in which the effects of a protocol of 12-week resistance training loading the Achilles tendon and low-energy focused extracorporeal shock wave therapy (ESWT) in patients with Achilles tendinopathy (AT) will be monitored. It is estimated that at least 40 patients will participate, randomly divided into two groups. Group A will be instructed to perform a training protocol in combination with ESWT according to selected parameters. Group B only completes the same training protocol.

DETAILED DESCRIPTION:
This work is designed as a randomized clinical trial, in which the effects of a protocol of 12-week resistance training loading the Achilles tendon and low-energy focused extracorporeal shock wave therapy (ESWT) in patients with Achilles tendinopathy (AT) will be monitored. It is estimated that at least 40 patients will participate, randomly divided into two groups. Group A will be instructed to perform a training protocol in combination with ESWT according to selected parameters. Group B only completes the same training protocol.

The research within one patient will last a total of 26 weeks from the initial to the final examination and will include several control measurements: at 6, 12, and 26 week from the beginning of therapy. Potential participants will be selected based on the recommendation of a specialist doctor and their suitability will be assessed according to the inclusion criteria. They will then be invited to an initial examination. This will include an objective examination by a physiotherapist, a subjective assessment by the patient and an ultrasonographic (USG) examination followed by a micromorphological analysis using special software. At the end of the initial examination, the participant will be randomly assigned to group A or B. The study program for a specific participant will depend on the assigned group.

ELIGIBILITY:
Inclusion Criteria:

* the patient shows symptoms of Achilles tendinopathy (pain, swelling and dysfunction in the area of Achilles tendon), which at least partially limit his quality of life during normal or sporting activities,
* the patient is in the age group of 18-60 years,
* the patient has difficulties in only one lower limb; the second, asymptomatic limb will be considered the reference,
* the patient is not aware of any mechanical damage to the tendon in symptomatic limb in the past (e.g. partial or complete rupture as a result of an injury),
* the patient has not undergone any treatment aimed at AS in the last 3 months (surgery, corticoid application, plasma therapy, shock waves, physiotherapy, etc.), objective US examination of AS shows structural changes (expansion, neovascularization, focal hypoechoic areas, etc.).

Exclusion Criteria:

* patient has been diagnosed with a rheumatic disease or a disease of the central nervous system
* patient has any condition which is contraindication for ESWT application
* patient is aware of mechanical damage to the Achilles tendon as a result of an injury in the past.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislav Machač, PhD, Study Chair — University Hospital Motol and 2nd Faculty of Medicine, Charles University
Locations (1):
- University Hospital Motol and 2nd Faculty of Medicine, Charles University, Prague, Czechia

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - ESWT + Exercise: Participants in group A will complete a 12-week ankle dorsiflexion resistance training protocol according to Silbernagel. It is a series of heel rise exercises with a gradual progression of load according to defined criteria, which the patient practices every day.
  In addition, participants will receive a low-energy focused ESWT. In total, it will be applied 4 times with an interval of 7 days from the BTL-6000 FSWT device with piezoelectric generator. The energy will be set to 0.10-0.14 mJ/mm2, frequency 6 Hz, total number of shocks 1800. The application will be semi-static at the location of the largest USG finding. 600 shocks are applied from all three sides (medial, lateral, dorsal). The set values will not change throughout the research. These parameters were selected in accordance to ISMST guidelines.
Period: Overall Study
Arm/Group | Group A - ESWT + Exercise | Group B - Exercise
Started | 23 | 24
Completed | 21 | 20
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Unrelated injury | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - ESWT + Exercise | Group B - Exercise | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (11.7) | 32.8 (11.8) | 33.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 14 | 11 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.7 (5.1) | 26.1 (4.4) | 24.9 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Peak Spatial Frequency Radius at the Site of Pathology
Description: Peak Spatial Frequency Radius (PSFR) was assessed using spatial frequency analysis (SFA) software applied to standardized B-mode ultrasound images of the Achilles tendon.
  Ultrasound images were acquired in a long-axis using predefined machine settings. The image was saved and exported for subsequent analysis. In the SFA software, the region corresponding to the site of maximal tendon pathology was selected, and PSFR values (mm-¹) were calculated.
  PSFR values were recorded at baseline and at the 26-week follow-up.
Time Frame: Values at baseline and week 26.
Measure: Mean (Standard Deviation); unit: mm^-1
Arm/Group | Group A - ESWT + Exercise | Group B - Exercise
Number analyzed (Participants) | 21 | 20
mm^-1
  Baseline | 2.180 (0.093) | 2.146 (0.067)
  Week 26 | 2.194 (0.115) | 2.184 (0.094)

2. Primary Outcome: VISA-A Questionnaire Score
Description: The VISA-A questionnaire is a validated, disease-specific patient-reported outcome measure for Achilles tendinopathy. Scores range from 0 to 100 (score on scale), with higher scores indicating better function and fewer symptoms.
  Scores were recorded at baseline and at the 26-week follow-up.
Time Frame: Values at baseline and week 26.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Group A - ESWT + Exercise | Group B - Exercise
Number analyzed (Participants) | 21 | 20
scores on scale
  Baseline | 66.9 (13.2) | 62.9 (12.8)
  Week 26 | 92.7 (7.2) | 86 (11.5)

3. Secondary Outcome: Tendon Diameter at the Place of Maximum Tendon Width
Description: Achilles tendon diameter was measured using standardized B-mode ultrasound imaging at the site of maximal tendon width. Measurements were performed using built-in ultrasound system measurement tools.
  Measurements were recorded at baseline and at the 26-week follow-up.
Time Frame: Values at baseline and week 26.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group A - ESWT + Exercise | Group B - Exercise
Number analyzed (Participants) | 21 | 20
mm
  Baseline | 6.0 (2.0) | 6.6 (2.2)
  Week 26 | 5.9 (1.9) | 6.4 (1.8)

4. Secondary Outcome: Pain Intensity Measured by Numeric Rating Scale (NRS)
Description: Pain intensity was assessed using an 11-point Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst imaginable pain).
  Scores were recorded at baseline and at the 26-week follow-up.
Time Frame: Values at baseline and week 26
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group A - ESWT + Exercise | Group B - Exercise
Number analyzed (Participants) | 21 | 20
scores on a scale
  Baseline | 6.8 (1.8) | 5.7 (1.6)
  Week 26 | 1.8 (1.4) | 1.9 (1.8)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 26 weeks
Description: No adverse effects (serious or others) were reported during treatment, after treatment and also during follow-up period.
Arm/Group | Group A - ESWT + Exercise | Group B - Exercise
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT05702918/Prot_SAP_000.pdf